CLINICAL TRIAL: NCT05174754
Title: The Impact Of A Physician-led Exercise Programme On Quality Of Life, Muscle Mass And Clinical Response In Inflammatory Bowel Disease Patients During Induction With Medical Therapy
Brief Title: Response To Medical Therapy in Inflammatory Bowel Disease Patients Carrying-out a Prescribed Exercise Programme
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-048
Record Dates: First submitted 2021-11-08; First posted 2022-01-03 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-02

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inflammatory Bowel Disease Exercise Group (Experimental): The exercise group will be randomized to a 20-week physician-prescribed exercise programme following the principles of Frequency, Intensity, Time, and Type (FITT) in addition to best medical therapy with the aim of increasing physical fitness levels, inflammatory response, quality of life/fatigue improvements and favorable body composition changes.
  Interventions: Behavioral: Physician-prescribed Exercise Programme; Drug: Best Medical Therapy
- Inflammatory Bowel Disease Control Group (Other): The IBD control group will be randomized to best medical therapy alone.
  Interventions: Drug: Best Medical Therapy
- Healthy Control Group (No Intervention): A group of healthy controls without inflammatory bowel disease will be included in the study for comparison of inflammatory markers including cytokine analysis and body composition.

INTERVENTIONS:
Behavioral: Physician-prescribed Exercise Programme — A 20-week structured exercise programme derived and supervised by a Sports Medicine Physician following the FITT Principles
  Arms: Inflammatory Bowel Disease Exercise Group
Drug: Best Medical Therapy — Best medical therapy with biologic agent or small-molecule therapy
  Arms: Inflammatory Bowel Disease Control Group; Inflammatory Bowel Disease Exercise Group

SUMMARY:
The investigators propose the use of a 20 week physician-derived exercise programme will lead to an improvement in physical fitness which will in turn lead to an increase in muscle mass, a reduction in visceral obesity resulting in an improvement in biologic response, disease biomarkers (including a reduction in circulating pro-inflammatory cytokines), fatigue scores and quality of life.

DETAILED DESCRIPTION:
After completion, the investigators expect to describe the significant impact that exercise has on IBD disease control, response to biologics, modification of pro-inflammatory cytokine levels, quality of life and fatigue scores.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or above.
* Confirmed moderate to severe inflammatory bowel disease based on endoscopic evaluation, clinical scoring tools and faecal calprotectin.
* Be able to provide written informed consent.
* Stable dose of steroids.
* Physically able to complete an exercise programme.
* Healthy controls.

Exclusion Criteria:

* Inability to participate in the exercise program (unable to perform 6MWT, unable to attend for assessment of parameters at any time point).
* An uncontrolled cardiovascular condition such as unstable angina, uncontrolled cardiac arrhythmias, uncontrolled symptomatic heart failure or symptomatic severe aortic stenosis.
* A significant musculoskeletal condition, neurological condition, mental illness or intellectual disability that restricts participation in a physical exercise program.
* Pregnancy.
* Healthy controls with underlying inflammatory conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-03-22 (Estimated); Study Completion 2023-05-22 (Estimated)

PRIMARY OUTCOMES:
The recruitment rates in both IBD arms. | 26 weeks
  A calculation of the percentage of people approached who participate in the intervention (recruitment).
The retention rate in both IBD arms. | 26 weeks
  A calculation of the percentage of people approached who complete the intervention.
The adherence rate in both IBD arms. | 26 weeks
  A calculation of the percentage of people approached who adhered to the intervention.

SECONDARY OUTCOMES:
Change in muscle mass measured by ultrasound | 26 weeks
  Ultrasound of thigh muscle mass (vastus intermedius and rectus femoris-measured in mm, subcutaneous adiposity measured in mm)
Change in muscle mass measured by bioelectrical impedance analysis | 26 weeks
  Bioelectrical impedance analysis (muscle mass in Kg)
Change in visceral fat measured by bioelectrical impedance analysis | 26 weeks
  Bioelectrical impedance analysis (visceral fat in Kg)
Clinical remission in response to exercise intervention | 12 and 26 weeks
  Harvey Bradshaw Index 2 or lower in Crohn's disease patients or partial Mayo score 0-1in ulcerative colitis
Change in fatigue score between the IBD groups in response to exercise | 12 and 26 weeks
  Measured using the Fatigue Severity Scale which comprises nine statements, describing the severity and impact of fatigue, with a scale of possible responses ranging from 1 ("strongly disagree") to 7 ("strongly agree").
Change in Quality of Life in response to exercise | 12 and 26 weeks
  Measured by the Short Inflammatory Bowel Disease Questionnaire (SIBDQ)- a ten item questionnaire, with 1 to 7 points for each item and higher scores indicating higher quality of life.
Change in endoscopic disease activity between IBD groups | 26 weeks
  A change in endoscopic appearance of Crohn's using Simple endoscopic score for Crohn's disease (SES CD) (inactive when SES-CD was 0-2; mild when 3-6; moderate 7-15; and severe >16) or Mayo score for ulcerative colitis (Score 0-3, Mayo 3 indicating severe disease, 2 moderate disease, 1 mild disease and 0 inactive).
Inflammatory response between IBD groups measured using C-Reactive protein | 12 and 26 weeks
  Change in C-Reactive Protein (mg/L)
Inflammatory response between IBD groups measured using faecal calprotectin | 12 and 26 weeks
  Change in faecal calprotectin (ug/g)
Inflammatory response between IBD groups measured using pro-inflammatory cytokines | 12 and 26 weeks
  Change in circulating pro-inflammatory cytokines (pg/mL)
Change in handgrip strength | 12 and 26 weeks
  Use of Jamar dynamometer to measure handgrip strength in kPa
A change in physical fitness between the IBD patient arms | 26 weeks
  15% difference in 6-minute walk test (6MWT) distance between the two groups

OTHER OUTCOMES:
Measurement of metabolic markers in response to exercise | 12 and 26 weeks
  Analysis of key immunometabolic pathways including flow cytometry of peripheral T-cells
Adverse events | 26 weeks
  The frequency and nature of adverse events will be recorded (number, percentage and type).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Boland, PhD, Principal Investigator — Royal College of Surgeons, Ireland and Beaumont Hospital, Dublin, Ireland.
Locations (1):
- Beaumont Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elia J, Kane S. Adult Inflammatory Bowel Disease, Physical Rehabilitation, and Structured Exercise. Inflamm Bowel Dis. 2018 Nov 29;24(12):2543-2549. doi: 10.1093/ibd/izy199. PMID 29850914
- [Background] Chan D, Robbins H, Rogers S, Clark S, Poullis A. Inflammatory bowel disease and exercise: results of a Crohn's and Colitis UK survey. Frontline Gastroenterol. 2014 Jan;5(1):44-48. doi: 10.1136/flgastro-2013-100339. Epub 2013 Jul 31. PMID 28839750
- [Background] Cronin O, Barton W, Moran C, Sheehan D, Whiston R, Nugent H, McCarthy Y, Molloy CB, O'Sullivan O, Cotter PD, Molloy MG, Shanahan F. Moderate-intensity aerobic and resistance exercise is safe and favorably influences body composition in patients with quiescent Inflammatory Bowel Disease: a randomized controlled cross-over trial. BMC Gastroenterol. 2019 Feb 12;19(1):29. doi: 10.1186/s12876-019-0952-x. PMID 30755154
- [Background] Eckert KG, Abbasi-Neureither I, Koppel M, Huber G. Structured physical activity interventions as a complementary therapy for patients with inflammatory bowel disease - a scoping review and practical implications. BMC Gastroenterol. 2019 Jul 2;19(1):115. doi: 10.1186/s12876-019-1034-9. PMID 31266461
- [Background] Gatt K, Schembri J, Katsanos KH, Christodoulou D, Karmiris K, Kopylov U, Pontas C, Koutroubakis IE, Foteinogiannopoulou K, Fabian A, Molnar T, Zammit D, Fragaki M, Balomenos D, Zingboim N, Ben Horin S, Mantzaris GJ, Ellul P. Inflammatory Bowel Disease [IBD] and Physical Activity: A Study on the Impact of Diagnosis on the Level of Exercise Amongst Patients With IBD. J Crohns Colitis. 2019 May 27;13(6):686-692. doi: 10.1093/ecco-jcc/jjy214. PMID 30561568
- [Background] Jones K, Baker K, Speight RA, Thompson NP, Tew GA. Randomised clinical trial: combined impact and resistance training in adults with stable Crohn's disease. Aliment Pharmacol Ther. 2020 Sep;52(6):964-975. doi: 10.1111/apt.16002. Epub 2020 Jul 30. PMID 33119156
- [Background] Jones PD, Kappelman MD, Martin CF, Chen W, Sandler RS, Long MD. Exercise decreases risk of future active disease in patients with inflammatory bowel disease in remission. Inflamm Bowel Dis. 2015 May;21(5):1063-71. doi: 10.1097/MIB.0000000000000333. PMID 25723616
- [Background] Klare P, Nigg J, Nold J, Haller B, Krug AB, Mair S, Thoeringer CK, Christle JW, Schmid RM, Halle M, Huber W. The impact of a ten-week physical exercise program on health-related quality of life in patients with inflammatory bowel disease: a prospective randomized controlled trial. Digestion. 2015;91(3):239-47. doi: 10.1159/000371795. Epub 2015 Mar 24. PMID 25823689
- [Background] Lamers CR, de Roos NM, Bongers CCWG, Ten Haaf DSM, Hartman YAW, Witteman BJM, Hopman MTE. Repeated prolonged moderate-intensity walking exercise does not appear to have harmful effects on inflammatory markers in patients with inflammatory bowel disease. Scand J Gastroenterol. 2021 Jan;56(1):30-37. doi: 10.1080/00365521.2020.1845791. Epub 2020 Nov 19. PMID 33211989
- [Background] Loudon CP, Corroll V, Butcher J, Rawsthorne P, Bernstein CN. The effects of physical exercise on patients with Crohn's disease. Am J Gastroenterol. 1999 Mar;94(3):697-703. doi: 10.1111/j.1572-0241.1999.00939.x. PMID 10086654
- [Background] Ng V, Millard W, Lebrun C, Howard J. Low-intensity exercise improves quality of life in patients with Crohn's disease. Clin J Sport Med. 2007 Sep;17(5):384-8. doi: 10.1097/JSM.0b013e31802b4fda. PMID 17873551
- [Background] Afzal R, Dowling JK, McCoy CE. Impact of Exercise on Immunometabolism in Multiple Sclerosis. J Clin Med. 2020 Sep 21;9(9):3038. doi: 10.3390/jcm9093038. PMID 32967206